CLINICAL TRIAL: NCT00912327
Title: A Phase 2 Efficacy and Safety, Open-label, Multicenter Study of Imprime PGG® Injection in Combination With Cetuximab in Subjects With Stage IV KRAS-Mutated Colorectal Cancer
Brief Title: Efficacy and Safety Study of Imprime PGG With Cetuximab in Subjects With Stage IV KRAS-Mutated Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: HiberCell, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BT-CL-PGG-CRC0821
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Colorectal Cancer
Keywords: Colorectal; KRAS mutation; Stage IV; Imprime PGG; Cetuximab; Immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue samples from previous biopsies and blood plasma will be collected.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Stage 1
  Interventions: Biological: Imprime PGG
- Stage 2
  Interventions: Biological: Imprime PGG

INTERVENTIONS:
Biological: Imprime PGG — Imprime PGG, 4 mg/kg, i.v. over 2 hr, weekly in 6 week cycles and Cetuximab, initial dose will be 400 mg/m2 via i.v., and subsequent doses will be 250 mg/m2 via i.v., weekly in 6 week cycles
  Other Names: Erbitux

SUMMARY:
Study BT-CL-PGG-CRC0821 is a Phase 2, open-label, multicenter, efficacy and safety study. It will be conducted using a two-stage design with the intention of determining the initial efficacy of Imprime PGG in combination with a monoclonal antibody (MAb; cetuximab) in the treatment of KRAS-mutant colorectal cancer (CRC). Both stages will be conducted in subjects with Stage IV CRC demonstrating the KRAS gene mutation. Subjects will dose until progression of disease or discontinuation from the study for other reasons; e.g., safety, non-compliance. Approximately 56 subjects will be enrolled at three participating centers (17 into Stage 1 and 39 into Stage 2).

DETAILED DESCRIPTION:
Study BT-CL-PGG-CRC0821 is a Phase 2, open-label, multicenter, efficacy and safety study. It will be conducted using a two-stage design with the intention of determining the initial efficacy of Imprime PGG in combination with a monoclonal antibody (MAb; cetuximab) in the treatment of KRAS-mutant colorectal cancer (CRC). Both stages will be conducted in subjects with Stage IV CRC demonstrating the KRAS gene mutation. All subjects will receive Imprime PGG at 4 mg/kg and standard doses of cetuximab; Imprime PGG and cetuximab will be administered in 6-week cycles. Subjects will dose until progression of disease or discontinuation from the study for other reasons; e.g., safety, non-compliance. The initial cetuximab dose will be 400 mg/m2 on Cycle 1/Day1 and subsequent doses of cetuximab will be 250 mg/m2 weekly. Imprime PGG will be dosed weekly at 4 mg/kg. Tumor measurements and determination of tumor responses for this study will be performed according to RECIST. Approximately 56 subjects will be enrolled at three participating centers (17 into Stage 1 and 39 into Stage 2). Final results will be determined from combined Stage 1 and Stage 2 data.

ELIGIBILITY:
Inclusion Criteria:

1. Is >18 years old;
2. Has Stage IV carcinoma of the colon or rectum with documented histological or cytological confirmation;
3. Tumor has known KRAS mutation;
4. Has failed previous irinotecan- and oxaliplatin-containing regimens in either adjuvant or metastatic settings or is intolerant to irinotecan-based therapies;
5. Has measurable disease, defined as at least one tumor that fulfills the criteria for a target lesion according to RECIST;
6. Has not received any other treatment for colorectal cancer within the 30 days prior to first dose of study treatment under this protocol;
7. Has an ECOG score of 0-1;
8. Has a life expectancy of > 3 months;
9. Has adequate bone marrow reserve as evidenced by:

   1. ANC ≥ 1,500/μL
   2. PLT ≥ 100,000/μL
10. Has adequate renal function as evidenced by serum creatinine ≤ 2.5X the upper limit of normal (ULN) for the reference lab;
11. Has adequate hepatic function as evidenced by:

    1. AST ≤ 3X ULN for the reference lab (≤ 5X ULN for subjects with known hepatic metastases)
    2. ALT ≤ 3X ULN for the reference lab (≤ 5X ULN for subjects with known hepatic metastases)
    3. Bilirubin < 1.5 mg/dl, OR direct bilirubin < 1.0 mg/dl
    4. Serum Albumin > 3.0 gm/dl
12. Has read, understood and signed the informed consent form (ICF) approved by the Independent Review Board/Ethics Committee (IRB/EC); and
13. If the subject is a woman of childbearing potential or a fertile man, he/she must agree to use an effective form of contraception during the study and for 60 days following the last dose of study medication (an effective form of contraception is abstinence, a hormonal contraceptive, or a double-barrier method).

Exclusion Criteria:

1. Has a known hypersensitivity to cetuximab, murine proteins, or any component of cetuximab;
2. Has a known hypersensitivity to baker's yeast or has an active yeast infection;
3. Has had previous exposure to Betafectin® or Imprime PGG;
4. Has an active, uncontrolled infection;
5. Has known or suspected brain metastases;
6. Had a second malignancy within the previous 5 years, except for basal cell carcinoma, cervical intra-epithelial neoplasia or curatively-treated prostate cancer with a PSA of < 2.0 ng/mL;
7. Has known HIV/AIDS, Hepatitis B, Hepatitis C, connective tissue disease, or other clinical diagnosis, ongoing or intercurrent illness that in the investigator's opinion should prevent participation;
8. If female, is pregnant or breast-feeding;
9. Is receiving concurrent standard and/or investigational anti-cancer therapy or has received such therapy within a period of 30 days prior to the first scheduled day of dosing (investigational therapy is defined as treatment for which there is currently no regulatory-authority-approved indication); or
10. Has previously received an organ or progenitor/stem cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 56 patients with Stage IV Kras-mutated colorectal cancer.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2009-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Assessed after 17 subjects complete 1 treatment cycle and at completion of study.

SECONDARY OUTCOMES:
Disease control rate (DCR) and duration of disease control | Assessed after 17 subjects complete 1 treatment cycle and at completion of study.
Complete response (CR), partial response (PR), and stable disease (SD) rates | Assessed after 17 subjects complete 1 treatment cycle and at completion of study.
Duration of objective tumor response | Assessed after 17 subjects complete 1 treatment cycle and at completion of study.
Duration of stable disease | Assessed after 17 subjects complete 1 treatment cycle and at completion of study.
Time to progression (TTP) | Assessed after 17 subjects complete 1 treatment cycle and at completion of study.
Progression-free survival (PFS) | Assessed after 17 subjects complete 1 treatment cycle and at completion of study.
Safety of the dosing regimen | Assessed after 17 subjects complete 1 treatment cycle and at completion of study.
Overall survival | Assessed after all subjects are deceased or lost to follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Saltz, MD, Principal Investigator — Memorial Sloane-Kettering Cancer Center; Neil H. Segal, MD, PhD, Principal Investigator — Memorial Sloane-Kettering Cancer Center; Neil Senzer, MD, Principal Investigator — Mary Crowley Medical Research Center; Purvi Gada, MD, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - University of Minnesota, Minneapolis, Minnesota
  - Memorial Sloane-Kettering Cancer Research Center, New York, New York
  - Mary Crowley Medical Research Center, Dallas, Texas